CLINICAL TRIAL: NCT00025311
Title: A Phase I Study Of Seven Day Continuous Intrathecal/Intraventricular Infusion Of Topotecan For Patients With Recurrent, Progressive Or Refractory Leptomingeal Disease
Brief Title: Topotecan in Treating Patients With Recurrent, Progressive, or Refractory Cancer That is Metastatic to the Lining Around the Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068949; NYU-0005H; NYU-0041H; NCI-G01-2018
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2003-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: leptomeningeal metastases
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningeal Carcinomatosis | interventions — Topotecan

INTERVENTIONS:
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of intrathecal or intraventricular topotecan in treating recurrent, progressive, or refractory cancer that is metastatic to the lining around the brain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of intrathecal or intraventricular topotecan in patients with recurrent, progressive, or refractory leptomeningeal disease.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine the anti-tumor activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to disease (leukemia or lymphoma vs solid tumor or other malignancy).

Patients receive topotecan intrathecally or intraventricularly continuously on days 1-7. Treatment repeats every 21 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose- limiting toxicity.

Patients are followed for 6 months.

PROJECTED ACCRUAL: A maximum of 50 patients (25 per stratum) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologic or tumor marker confirmation of malignancy at original diagnosis
* Neoplastic meningitis/leptomeningeal metastasis refractory to conventional therapy and other therapies of higher priority, defined as:

  * Stratum A:

    * Small non-cleaved lymphoma (Burkitt's) with any L-3 blast in cerebrospinal fluid (CSF)
    * Any other lymphoma or leukemia with CSF cell count greater than 5/mm3 AND evidence of blast cells by cytology or cytospin preparation OR
  * Stratum B:

    * Solid tumor or other malignancy with presence of tumor cells on cytospin OR positive cytology OR neuroimaging evidence of leptomeningeal tumor by MRI or CT myelogram
* No leptomeningeal leukemia or lymphoma with concurrent bone marrow relapse
* No clinical evidence of untreated obstructive hydrocephalus or compartmentalization of the CSF

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* Lansky 50-100% (age 16 and under)
* Karnofsky 50-100% OR ECOG 0-3 (over age 16)

Life expectancy:

* At least 2 months

Hematopoietic:

* Stratum B:

  * Absolute neutrophil count at least 750/mm^3
  * Platelet count at least 75,000/mm^3 (transfusion independent)
  * Hemoglobin at least 10.0 g/dL (red blood cell transfusions allowed)

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT or SGPT less than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Neurologic:

* Seizures allowed if well controlled and on anticonvulsants
* CNS toxicity no greater than grade 2

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infections
* HIV allowed

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunomodulating agents (stratum B)
* No stem cell transplantation (stratum A)

Chemotherapy:

* At least 2 weeks since prior chemotherapy (4 weeks for nitrosoureas)
* No other concurrent cancer chemotherapy (stratum B)
* Other concurrent systemic cancer chemotherapy for leukemia or lymphoma allowed with the following restrictions:

  * No oral or IV topotecan
  * No moderate or high-dose IV or subcutaneous cytarabine (greater than 1.0 g/m2 per day)
  * No moderate or high-dose IV methotrexate (greater than 1 g/m2 per day)
  * No IV thiotepa
  * No myeloablative chemotherapy
  * No intrathecal or intraventricular chemotherapy

Endocrine therapy:

* Concurrent corticosteroids allowed only for treatment of increased intracranial pressure in patients with CNS tumors
* No concurrent intrathecal or intraventricular hydrocortisone

Radiotherapy:

* At least 4 weeks since completion of radiotherapy to the brain or spine and recovered
* Concurrent radiotherapy to localized painful lesions producing acute neurologic dysfunction allowed provided at least 1 measurable lesion is not irradiated
* No concurrent craniospinal or whole-brain radiotherapy

Surgery:

* Not specified

Other:

* Recovered from prior therapy
* At least 7 days since prior investigational drug
* No other concurrent intrathecal or intraventricular therapy for leptomeningeal disease

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-05; Primary Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan L. Finlay, MB, ChB, Study Chair — NYU Langone Health
Locations (3):
- United States (2):
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
- CHU Pitie-Salpetriere, Paris, France